CLINICAL TRIAL: NCT06341738
Title: The Efficacy of Digital Educational Interventions on Parental HPV Knowledge and Attitude, and Their Children's HPV Vaccination Rates in Indonesia
Brief Title: The Efficacy of Digital Educational Interventions on Parental HPV Knowledge and Attitude, and Their Children's Vaccination Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Yudisa Diaz Lutfi Sandi, RN., MSN., PhD Candidate (Principal Investigator), Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 421/215/404.102.28/VI/2023
Record Dates: First submitted 2024-03-15; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Health Services Research
Keywords: vaccine; human papillomavirus; digital education; parent; trial
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Intervention Model Description: 10 units are divided into 2 arms (e.g. intervention and control) by cluster randomisation using the number of units into a sealed envelope. the participants are unaware of which group they were placed in
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIgital Education Group (Experimental): The intervention group will receive information on HPV and the HPV vaccine from an 8-minute video in front of the class, two electronic reminder messages send to participant before the vaccination events
  Interventions: Behavioral: Video education about HPV and HPV vaccine; Behavioral: Electronic reminder messages
- Usual Information Service Group (Active Comparator): the control group will only receive the usual information service from staff
  Interventions: Behavioral: Usual Information Service

INTERVENTIONS:
Behavioral: Video education about HPV and HPV vaccine — video animation in 8 minutes to promote about HPV and HPV vaccine. the video is played in front of class using LCD projector.
  Arms: DIgital Education Group
Behavioral: Electronic reminder messages — Reseachers send reminder messages twice per vaccination event (e.g., 7 days and 1 day before vaccination event), with a total of four times sending reminder messages using the app on the smartphone.
  Arms: DIgital Education Group
Behavioral: Usual Information Service — this usual information (e.g., the HPV vaccination event) was delivered face-to-face by staff in front of class
  Arms: Usual Information Service Group

SUMMARY:
The goal of this clinical trial is to examine in the parental HPV knowledge and attitude, and their children's completion rates in Indonesia. The main question[s] it aims to answer are:

* Is the digital educational intervention in improving parent's HPV knowledge in the intervention group compared to the control group?
* Is the digital educational intervention in improving parent's attitude toward HPV vaccine in the intervention group compared to the control group?
* Is the digital educational intervention more effective in increasing children's HPV vaccine completion rates in the intervention group compared to the control group?

Participants in intervention group will:

* watch a 8 minutes video in front of class at once.
* after video education intervention, in 2 weeks, participants received 2 reminder messages before first and second vaccination event, respectively.

Participants in control group will:

• Receive usual announcement regarding vaccine by staff

DETAILED DESCRIPTION:
Research process started after obtaining permission principal of the elementary school and primary health centre. Because the target population was parents of girls in the 5-6th level, permission was required from the elementary schools. Meanwhile, another permission must be obtained from the Primary Health Centre, they have authority to administer the HPV vaccine to children at the school.

All participants (parents) were recruited from 10 elementary schools. The schools were divided into 2 arm (e.g., Digital education group, Usual information service group) by cluster randomizing. The group allocation were concealed from the participants, elementary teachers and primary health centre. Participants were unaware of the existence of any other group than the one they received. According to sample size calculations, the number of adequate sample sizes in this study based on sample size calculation results at the completion rate. The dropout rate estimation of 10% according to a previous study by Reiter (2022), the total sample size increased to 269 + (10% x 269) = 296 participants.

The researchers got an approval from schools to invite parents to attend the school of event invitations. Each participant came to the school where their child attended. Parents attended the regular meeting on the appointed day. Frequently, event invitations have become a routine program in elementary school. It was a routine agenda to socialize interesting programs related to students and parents. In parallel with the above, the research team coordinated with the Primary Health Center as the administrator of the HPV vaccine in elementary schools. Thus, the research team determined the time to give the digital education intervention and the follow-up evaluation.

During the process, the researchers approached potential participants and explain to them the purpose of this study, participant rights, risks, and benefits. Then potential participants were asked to sign in the informed consent form with serial numbel. The outcome measurement questionnaires were distributed to the participants, either the intervention group or the control group.

At baseline, the eligible participants were asked to fill out the questionnaires. After complete, a 8 minutes video was played in front of class. Then, the participants took a post-test right after the intervention finish their meeting and in the control group as well. The post-test assessed HPV knowledge and attitudes toward the HPV vaccine. Prior vaccination events, the reminder messages were sent to parent's mobile phone. At this stage, the researcher observed the first dose of HPV vaccine uptake among female students during the HPV vaccine administration program at school. The researcher collected data by observing female students who received the first and second doses of HPV vaccine at the vaccination event, then confirmed the researcher's observations with the Primary Health Center record. All data was recapitulated and stored in excel format. Data was kept by the researcher to maintain confidentiality. All data analyses were performed using SPSS software from IBM Corp.

Statistical analyses, below:

1. Pearson Chi-Square test or Fisher's exact test was used to analyse the HPV vaccine completion rate between groups.
2. The T-test was used to analyse the HPV knowledge and attitude towards HPV vaccine between groups;
3. ANCOVA analysed the intervention efficacy on knowledge, attitude, and HPV vaccine completion rate between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Parents over 17 years old
* Parents Parents who have daughters of 5-6th level in elementary school
* Parents live with their children in one house
* Parents have a mobile phone with WhatsApp application capabilities
* Parents who have their daughters have been enrolled in School-Based Immunization Program database
* Parents able to communicate fluently in Bahasa Indonesia
* Parents agree to review their child's medical record of vaccination

Exclusion Criteria:

* Parents have diagnosed with mental, visual, and hearing impairment/problems diagnosed by doctors
* Parents whose children have been HPV vaccinated
* Parents whose children are over 14 years old
* Children who have a history of allergies and/or side effects in previous vaccination programs

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Human Papillomavirus Knowledge Scale (HPV-KS) | measured at pre-test/baseline (before the 8-minutes video) and post-test (immediately after watching the 8-minutes video).
  consist of 33 items divided into 3 factors with binary respond format (true/false). the correct answer indicated "1" point. The sum of items is HPV knowledge level. High score indicated high knowledge about HPV
Attitude towards HPV vaccine scale by Carolina HPV Immunization Attitudes and Beliefs Scale (CHIAS) | measured at pre-test/baseline (before the 8-minutes video) and post-test (immediately after watching the 8-minutes video).
  consist of 14 items divided into 3 factors with 4-Likert scale. A high mean score total attitude indicated a high positive attitudes
Vaccine completion rate | The evaluation was conducted twice, at week 2 post video intervention or at first vaccination event and 6 months later at second vaccination event.
  Receipt of two doses is considered vaccine series completion according vaccine policy in Indonesia

CONTACTS AND LOCATIONS:
Overall Officials: Yudisa Diaz Lutfi Sandi, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Elementary school, Ngawi, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
due to confidentiality protocols, participant data cannot be shared.

REFERENCES:
- [Result] Chen H, Zhang X, Wang W, Zhang R, Du M, Shan L, Li Y, Wang X, Liu Y, Zhang W, Li X, Qiao Y, Ma J, Zhou J, Li J. Effect of an educational intervention on human papillomavirus (HPV) knowledge and attitudes towards HPV vaccines among healthcare workers (HCWs) in Western China. Hum Vaccin Immunother. 2021 Feb 1;17(2):443-450. doi: 10.1080/21645515.2020.1780093. Epub 2020 Jul 21. PMID 32692948
- [Result] Chao C, Preciado M, Slezak J, Xu L. A randomized intervention of reminder letter for human papillomavirus vaccine series completion. J Adolesc Health. 2015 Jan;56(1):85-90. doi: 10.1016/j.jadohealth.2014.08.014. Epub 2014 Nov 1. PMID 25438965
- [Result] Bruni L, Diaz M, Barrionuevo-Rosas L, Herrero R, Bray F, Bosch FX, de Sanjose S, Castellsague X. Global estimates of human papillomavirus vaccination coverage by region and income level: a pooled analysis. Lancet Glob Health. 2016 Jul;4(7):e453-63. doi: 10.1016/S2214-109X(16)30099-7. PMID 27340003
- [Result] Wynn CS, Catallozzi M, Kolff CA, Holleran S, Meyer D, Ramakrishnan R, Stockwell MS. Personalized Reminders for Immunization Using Short Messaging Systems to Improve Human Papillomavirus Vaccination Series Completion: Parallel-Group Randomized Trial. JMIR Mhealth Uhealth. 2021 Dec 27;9(12):e26356. doi: 10.2196/26356. PMID 34958306
- [Result] Taebi M, Riazi H, Keshavarz Z, Afrakhteh M. Knowledge and Attitude Toward Human Papillomavirus and HPV Vaccination in Iranian Population: A Systematic Review. Asian Pac J Cancer Prev. 2019 Jul 1;20(7):1945-1949. doi: 10.31557/APJCP.2019.20.7.1945. PMID 31350949
- [Result] Szilagyi PG, Schaffer S, Shone L, Barth R, Humiston SG, Sandler M, Rodewald LE. Reducing geographic, racial, and ethnic disparities in childhood immunization rates by using reminder/recall interventions in urban primary care practices. Pediatrics. 2002 Nov;110(5):e58. doi: 10.1542/peds.110.5.e58. PMID 12415064
- [Result] Santhanes D, Yong CP, Yap YY, Saw PS, Chaiyakunapruk N, Khan TM. Factors influencing intention to obtain the HPV vaccine in South East Asian and Western Pacific regions: A systematic review and meta-analysis. Sci Rep. 2018 Feb 26;8(1):3640. doi: 10.1038/s41598-018-21912-x. PMID 29483541
- [Result] Rodriguez AM, Do TQN, Goodman M, Schmeler KM, Kaul S, Kuo YF. Human Papillomavirus Vaccine Interventions in the U.S.: A Systematic Review and Meta-analysis. Am J Prev Med. 2019 Apr;56(4):591-602. doi: 10.1016/j.amepre.2018.10.033. Epub 2019 Feb 15. PMID 30773231
- [Result] Pot M, Paulussen TG, Ruiter RA, Eekhout I, de Melker HE, Spoelstra ME, van Keulen HM. Effectiveness of a Web-Based Tailored Intervention With Virtual Assistants Promoting the Acceptability of HPV Vaccination Among Mothers of Invited Girls: Randomized Controlled Trial. J Med Internet Res. 2017 Sep 6;19(9):e312. doi: 10.2196/jmir.7449. PMID 28877862
- [Result] Ortiz RR, Smith A, Coyne-Beasley T. A systematic literature review to examine the potential for social media to impact HPV vaccine uptake and awareness, knowledge, and attitudes about HPV and HPV vaccination. Hum Vaccin Immunother. 2019;15(7-8):1465-1475. doi: 10.1080/21645515.2019.1581543. Epub 2019 Apr 11. PMID 30779682
- [Result] McCann L, McMillan KA, Pugh G. Digital Interventions to Support Adolescents and Young Adults With Cancer: Systematic Review. JMIR Cancer. 2019 Jul 31;5(2):e12071. doi: 10.2196/12071. PMID 31368438
- [Result] Magaard JL, Seeralan T, Schulz H, Brutt AL. Factors associated with help-seeking behaviour among individuals with major depression: A systematic review. PLoS One. 2017 May 11;12(5):e0176730. doi: 10.1371/journal.pone.0176730. eCollection 2017. PMID 28493904
- [Result] Lu B, Kumar A, Castellsague X, Giuliano AR. Efficacy and safety of prophylactic vaccines against cervical HPV infection and diseases among women: a systematic review & meta-analysis. BMC Infect Dis. 2011 Jan 12;11:13. doi: 10.1186/1471-2334-11-13. PMID 21226933
- [Result] Lopez N, Garces-Sanchez M, Panizo MB, de la Cueva IS, Artes MT, Ramos B, Cotarelo M. HPV knowledge and vaccine acceptance among European adolescents and their parents: a systematic literature review. Public Health Rev. 2020 May 14;41:10. doi: 10.1186/s40985-020-00126-5. eCollection 2020. PMID 32435520
- [Result] Loke AY, Kwan ML, Wong YT, Wong AKY. The Uptake of Human Papillomavirus Vaccination and Its Associated Factors Among Adolescents: A Systematic Review. J Prim Care Community Health. 2017 Oct;8(4):349-362. doi: 10.1177/2150131917742299. Epub 2017 Nov 21. PMID 29161946
- [Result] Dorji T, Nopsopon T, Tamang ST, Pongpirul K. Human papillomavirus vaccination uptake in low-and middle-income countries: a meta-analysis. EClinicalMedicine. 2021 Apr 17;34:100836. doi: 10.1016/j.eclinm.2021.100836. eCollection 2021 Apr. PMID 33997733
- [Result] Tudor Car L, Soong A, Kyaw BM, Chua KL, Low-Beer N, Majeed A. Health professions digital education on clinical practice guidelines: a systematic review by Digital Health Education collaboration. BMC Med. 2019 Jul 18;17(1):139. doi: 10.1186/s12916-019-1370-1. PMID 31315642